CLINICAL TRIAL: NCT03328078
Title: An Open-Label, Dose Escalation and Dose Expansion Trial Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Orally Administered CA-4948 in Patients With Relapsed or Refractory Primary Central Nervous System Lymphoma
Brief Title: CA-4948-101: Open-Label, Dose Escalation and Expansion Trial of Emavusertib (CA-4948) in Relapsed or Refractory Primary Central Nervous System Lymphoma (R/R PCNSL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA-4948-101; 2024-513312-95-00 (EU CTIS Number); 2022-000891-20 (EudraCT Number)
Record Dates: First submitted 2017-10-17; First posted 2017-11-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Relapsed Hematologic Malignancy; Refractory Hematologic Malignancy; Relapsed Primary Central Nervous System Lymphoma; Refractory Primary Central Nervous System Lymphoma
Keywords: MYD88; IRAK4; NHL; PCNSL; Lymphoma; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Relapsed/refractory Central Nervous System (CNS) Lymphoma; Systemic Lymphoma with Concurrent CNS Lymphoma; Systemic Lymphoma with a History of Treated CNS Lymphoma; Ibrutinib; Bruton tyrosine kinase inhibitor (BTKi); Primary CNS Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Recurrence | interventions — CA-4948; ibrutinib

STUDY DESIGN:
Intervention Model Description: Part A will evaluate escalating doses of emavusertib (CA-4948) either as monotherapy (Part A1) or in combination with ibrutinib (Part A2). Enrollment is closed for Part A1 and A2. Part B will comprise two expansion cohorts to assess efficacy and safety of emavusertib in combination with ibrutinib in R/R PCNSL. Part C will comprise three cohorts to assess the efficacy and safety of emavusertib monotherapy, ibrutinib monotherapy, and emavusertib in combination with ibrutinib in participants with R/R PCNSL who are naïve to BTKi treatment.
Masking Description: Part B is non-randomized and Part C is randomized.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Emavusertib (CA-4948) dose escalation (Experimental): Part A1: Dose-level cohorts with up to approximately 6 participants each will be used to define the Maximum Tolerated Dose (MTD) for emavusertib.
  Interventions: Drug: Emavusertib
- Emavusertib (CA-4948) and ibrutinib dose escalation (Experimental): Part A2: Evaluate escalating dose levels of oral emavusertib in combination with 560 mg QD or 420 mg QD of oral ibrutinib. The starting dose of emavusertib to be used in combination will be 200 mg BID. It is anticipated that 12 to 20 participants at a potential dose level will be required to establish optimal combination dosing.
  Interventions: Drug: Emavusertib; Drug: Ibrutinib
- Emavusertib (CA-4948) and ibrutinib dose expansion (Experimental): In two Expansion Cohorts (Part B), emavusertib in combination with ibrutinib will be administered in participants with R/R PCNSL who have progressed on a BTKi. In Cohort 1, emavusertib 100 mg BID will be administered with ibrutinib 560 mg QD consecutively in 28-day treatment cycles. In Cohort 2, emavusertib 200 mg BID will be administered with ibrutinib 560 mg QD consecutively in 28-day treatment cycles.
  Interventions: Drug: Emavusertib; Drug: Ibrutinib
- Emavusertib (CA-4948) and ibrutinib (Experimental): In this part of the study (Part C), eligible second-line participants with R/R PCNSL who are naïve to BTKi treatment will receive 1 of 3 treatment arms: (1) emavusertib 200 mg BID, (2) ibrutinib 560 mg QD, or (3) emavusertib 200 mg BID in combination with ibrutinib 560 mg QD. Treatments will be administered continuously in 28-day treatment cycles.
  Interventions: Drug: Emavusertib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Emavusertib — Emavusertib will be provided as a tablet dosage form to be taken BID.
  Other Names: CA-4948
Drug: Ibrutinib — Ibrutinib will be provided as a tablet or capsule dosage form to be taken QD.
  Arms: Emavusertib (CA-4948) and ibrutinib; Emavusertib (CA-4948) and ibrutinib dose escalation; Emavusertib (CA-4948) and ibrutinib dose expansion

SUMMARY:
This is a multi-center, open-label study to evaluate the safety, pharmacokinetics (PK), and anti-cancer activity of oral administration of emavusertib alone or in combination with ibrutinib in adult participants with relapsed or refractory (R/R) hematologic malignancies.

This trial will be completed in four parts. In Part A1, emavusertib will be evaluated first in a dose escalating monotherapy setting to establish the safety and tolerability (complete). In Part A2, emavusertib will be evaluated in combination with ibrutinib at 560 milligrams (mg) once daily (QD) or 420 mg QD as indicated by disease (Part A2 complete).

Part B will comprise 2 cohorts to assess safety and efficacy of emavusertib in combination with ibrutinib in participants with R/R primary central nervous system lymphoma (PCNSL) who have directly progressed on a bruton tyrosine kinase inhibitor (BTKi). In this part of the study, emavusertib will be dosed at 100 mg or 200 mg twice daily (BID) in combination with ibrutinib in 28-day treatment cycles.

Part C will comprise 3 treatment arms in the second-line setting to assess the efficacy and safety of emavusertib monotherapy, ibrutinib monotherapy, and emavusertib in combination with ibrutinib in participants with R/R PCNSL who are naïve to BTKi treatment. In this part of the study, eligible second-line participants with R/R PCNSL who are naïve to BTKi treatment will be randomized 1:1:1 to 1 of 3 treatment arms: (1) emavusertib 200 mg BID, (2) ibrutinib 560 mg QD, or (3) emavusertib 200 mg BID in combination with ibrutinib 560 mg QD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females greater than or equal to 18 years of age
2. Life expectancy of at least 3 months
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
4. Histopathologically confirmed diagnosis of PCNSL (medical record is acceptable). Cerebral biopsies are not required if imaging reveals typical images of PCNSL.

   1. Participants with parenchymal lesions must have unequivocal evidence of disease progression (e.g., presence of at least 1 measurable target lesion [≥ 10 millimeters (mm) and ≤ 40 mm in the longest diameter on brain magnetic resonance imaging [MRI] or head computed tomography [CT] on imaging within 28 days prior to Cycle 1 Day 1]). In cases where the tumor size is smaller but still measurable and located at a critical central nervous system (CNS) location, disabling the participant and/or causing symptoms, this participant may be eligible following a discussion with the Sponsor Medical Monitor.
   2. For participants limited to leptomeningeal involvement, cerebrospinal fluid (CSF) analysis (cytology and/or flow cytometry) with or without additional imaging (MRI) of the spine as clinically indicated is required to document abnormal cells within 28 days prior to Cycle 1 Day 1.

Exclusion Criteria for Part B and Part C

1. Participants with only intraocular PCNSL without brain lesion or CSF involvement, T-cell lymphoma, systemic presence of lymphoma, or non-CNS lymphoma metastatic to the CNS
2. Evidence of systemic lymphoma. This must be demonstrated by a positron emission tomography (PET) scan (or CT scan with contrast if applicable) of the chest, abdomen, and pelvis at Screening (testicular ultrasound may be considered to exclude a testicular lymphoma disseminated to the brain).
3. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) or prior history of systemic lymphoma, unless the participant has been free of the disease for ≥ 3 years.
4. Active malignancy other than PCNSL requiring systemic therapy
5. Previous BTKi treatment (Part C only).
6. History of Grade ≥ 3 rhabdomyolysis without complete recovery
7. Requirement for urgent therapy due to uncontrolled tumor mass/edema effects.
8. Received external beam radiation therapy to the CNS within 28 days prior to Cycle 1 Day 1.
9. Received prior investigational drugs (including treatment in clinical research, unapproved combination products, and new dosage forms) within 28 days or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1; allogeneic hematopoietic stem cell transplant (HSCT) within 60 days prior to Cycle 1 Day 1; or had clinically significant graft-versus-host disease (GVHD) requiring ongoing up-titration of immunosuppressive medications prior to Screening (with the exception of a BTKi for Part B only).

   Note: The use of a stable or tapering dose of immunosuppressive therapy post-HSCT and/or topical steroids for ongoing skin GVHD is permitted with Sponsor Medical Monitor approval
10. Any prior systemic anti-cancer treatment such as chemotherapy, immunomodulatory drug therapy, etc., received within 14 days or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1 (with the exception of ibrutinib or other BTKi for Part B only, which may be continued until the day before Cycle 1 Day 1)
11. Prior history of hypersensitivity or anaphylaxis to emavusertib, ibrutinib or any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Part A: To determine the safety and tolerability of emavusertib as a monotherapy and in combination with ibrutinib: dose-limiting toxicity (DLT) | 12 months
  The number of participants with a dose-limiting toxicity (DLT) in the first treatment cycle
Part A: Maximum tolerated dose (MTD) of emavusertib as a monotherapy and in combination with ibrutinib measured by dose-limiting toxicities (DLTs) | 12 months
  MTD determined by the highest dose level studied at which fewer than 2 out of 6 subjects (<33%) experience a dose limiting toxicity.
Part A: Recommended Phase 2 Dose (RP2D) of emavusertib as a monotherapy and in combination with ibrutinib based on overall tolerability data | 12 months
  RP2D selected based on overall tolerability data from all participants treated at different dose levels and will not exceed the MTD.
Part B: Overall Response Rate (ORR) in participants with R/R PCNSL | 18 months
Part C: ORR in participants with R/R PCNSL | 18 months

SECONDARY OUTCOMES:
Parts A, B and C: Pharmacokinetic (PK) profile of emavusertib and ibrutinib measured by AUC | 24- 66 months
  Area Under the concentration-time curve (AUC)
Parts A, B and C: Pharmacokinetic (PK) profile of emavusertib and ibrutinib measured by Cmax | 24- 66 months
  Maximum plasma concentration (Cmax)
Parts A, B and C: Pharmacokinetic (PK) profile of emavusertib and ibrutinib measured by Cmin | 24- 66 months
  Minimum plasma concentration (Cmin)
Parts A, B and C: Pharmacokinetic (PK) profile of emavusertib and ibrutinib measured by Tmax | 24- 66 months
  Time to maximum plasma concentration (Tmax)
Parts A, B and C: Pharmacokinetic (PK) profile of emavusertib and ibrutinib measured by plasma terminal half-life | 24- 66 months
  Plasma terminal elimination half-life (T 1/2)
Part A: To assess efficacy of emavusertib as a monotherapy and in combination with ibrutinib measured by ORR | 24- 36 months
  Assessed by ORR
Parts A, B and C: To assess efficacy of emavusertib as a monotherapy and in combination with ibrutinib and ibrutinib as monotherapy measured by duration of response (DOR) | 24- 66 months
  Assessed by DOR
Part A: To assess efficacy of emavusertib as a monotherapy and in combination with ibrutinib measured by disease control rate (DCR) | 24- 36 months
  Assessed by DCR
Parts A, B and C: To assess efficacy of emavusertib as a monotherapy and in combination with ibrutinib and ibrutinib as monotherapy measured by progression free survival (PFS) | 24- 66 months
  Assessed by PFS
Parts A, B and C: To assess efficacy of emavusertib as a monotherapy, in combination with ibrutinib and ibrutinib as monotherapy measured by overall survival (OS) | 24 - 66 months
  Assessed by OS
Parts B and C: To assess the safety and tolerability of emavusertib as monotherapy, ibrutinib as monotherapy and emavusertib in combination with ibrutinib in participants with R/R PCNSL | up to 66 months
  Measured by the number of participants with treatment-emergent adverse events (TEAEs) and treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (43):
- United States (27):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Providence St. John's Health Center, Santa Monica, California
  - UCLA Department of Medicine - Hematology/Oncology, Santa Monica, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Fred and Pamela Buffett Cancer Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Mt Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Duke Cancer Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Neurological Specialties West, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Hilman Cancer Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- France (4):
  - Institut Bergonie, Bordeaux
  - Hopital de la Timone, Marseille
  - Hospital Pitie Salpetriere, Paris
  - Institut Curie Hospital, Paris
- Israel (2):
  - Hematology Department Soroka UMC / Heanatology Department, Beersheba
  - Hadassah Medical Center / Ein-Carem, Jerusalem
- Italy (4):
  - Università di Torino Croce e Carle, Cuneo
  - SODc Ematologia Azienda Ospedaliera Universitaria Careggi, Florence
  - IRST - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS San Raffaele Scientific Institute, Milan
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne Osrodek Badan Klinicznych Wczesnych Faz, Gdansk
  - Oddzial Kliniczny Hematologii, Krakow
  - NarodowyInstytutu Onkologii im. Marii Sklodowskiej-Curie-Panstwowy Instytutu Badawczy, Warsaw
- Spain (2):
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen del Rocio, Seville